CLINICAL TRIAL: NCT01937039
Title: Johns Hopkins Breast Cancer Program Longitudinal Repository
Status: Active, not recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: J0888; SKCCC J0888 (Other: SKCCC at Johns Hopkins); NA_00019811 (Other: JHM IRB)
Record Dates: First submitted 2013-09-03; First posted 2013-09-09 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Benign Breast Disease
MeSH Terms: conditions — Breast Neoplasms; Cystic Fibrosis | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for example: whole blood, serum, plasma, urine, and tissue samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Breast cancer patients: Participants have a known diagnosis of breast cancer and are receiving a breast cancer evaluation and/or treatment, who agree to sample collection, access, and follow-up as part of the repository.
  Interventions: Procedure: Sample collection
- Benign breast disease: Participants have benign breast disease and are receiving a diagnostic procedure and/or evaluation, who agree to sample collection, access, and follow-up as part of the repository.
  Interventions: Procedure: Sample collection
- Healthy volunteer: Participants have no known diagnosis of breast disease or abnormality and are undergoing routine screening or diagnostic breast imaging procedures and/or other clinical evaluation, who agree to sample collection, access, and follow-up as part of the repository.
  Interventions: Procedure: Sample collection

INTERVENTIONS:
Procedure: Sample collection — Blood, tissue, urine, and other samples may be collected

SUMMARY:
The Breast Cancer Program Longitudinal Repository (BCPLR) is being established to fulfill the research mission of the Breast Cancer Program at Johns Hopkins and to serve investigators affiliated with it - to develop a repository of specimens with corresponding characteristics from patients seen in the breast care and cancer clinics.

DETAILED DESCRIPTION:
This research is being done to collect samples for future use that we may learn more about cancer by studying cells in blood and tissue collected from people with breast cancer as well as from volunteers without breast cancer. Our goal is to make these available for research to help to learn how cancer develops and how it may be treated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Participants meet one of the following categories: have a known diagnosis of breast cancer receiving a breast cancer evaluation and/or treatment; have benign breast disease receiving a diagnostic procedure and/or evaluation; or, have no known diagnosis of breast disease or abnormality and is undergoing routine screening or diagnostic breast imaging procedures and/or other clinical evaluation.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any man or woman being seen at Johns Hopkins for breast cancer treatment, or for any screening or diagnostic breast procedures (for example: mammograms or biopsies), may join. Individuals without a history of breast cancer, known as "healthy" or "normal" volunteers (meaning they do not have breast cancer) may also join.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Actual)
Dates: Start 2009-04; Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Repository development | 20 years
  To develop a repository of specimens with corresponding characteristics - demographic and clinical information - from patients seen in the breast care and cancer clinics

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. Wolff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States